CLINICAL TRIAL: NCT05505344
Title: Exploring the Validity of Seismofit® for Estimating Peak Oxygen Uptake in People With Coronary Heart Disease
Brief Title: Estimating Peak Oxygen Uptake in People Living With Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other); Northumbria University (Other); VentriJect ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: ER45328094
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation lab study: All participants will have a resting and exercising electrocardiogram (ECG) trace and a lung function test, called spirometry, will be performed. They will take part in a maximal CPET to determine V̇O2 peak. Participants will also have their V̇O2 peak estimated twice, twenty minutes apart, using the VentriJect Seismofit device. A short questionnaire will be administered to explore the acceptability of completing a maximal CPET and having V̇O2 peak estimated using VentriJect Seismofit.
  Interventions: Device: VentriJect Seismofit validation

INTERVENTIONS:
Device: VentriJect Seismofit validation — All participants will have a resting and exercising electrocardiogram (ECG) trace and a lung function test, called spirometry, will be performed. They will take part in a maximal CPET to determine V̇O2 peak. Participants will also have their V̇O2 peak estimated twice, twenty minutes apart, using the VentriJect Seismofit device. A short questionnaire will be administered to explore the acceptability of completing a maximal CPET and having V̇O2 peak estimated using VentriJect Seismofit.

SUMMARY:
In people living with coronary heart disease (CHD), V̇O2 peak predicts all-cause mortality. V̇O2 peak increases with regular exercise training. Thus, in exercise-based cardiovascular rehabilitation programmes, V̇O2 peak is a useful marker of how effective the exercise training has been.

Maximal cardiopulmonary exercise testing (CPET) is the gold standard method of measuring V̇O2 peak. However, maximal CPET is expensive and requires trained staff to conduct the test and interpret the results. Furthermore, CPET is not routinely available in United Kingdom (UK) cardiovascular rehabilitation programmes. Field exercise tests, such as incremental cycle ergometer tests, are used in conjunction with predictive equations to estimate V̇O2 peak. However, this group has shown that estimating changes in V̇O2 peak in this way is inaccurate. Alternative solutions are required.

VentriJect Seismofit® uses a technique called seismocardiography (SCG); the measurement of vibrations in the chest wall, caused by each heartbeat, using accelerometers. SCG can be used to estimate V̇O2 peak from a SCG measurement taken at rest. This study will explore the validity of VentriJect Seismofit for estimating V̇O2 peak in people with CHD.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary heart disease
* Able to lay fully supine for five minutes
* Capable of performing a maximum effort CPET on a stationary cycle ergometer
* Currently enrolled in a Phase IV cardiac rehabilitation programme
* A minimum of 12 weeks after a cardiac event

Exclusion Criteria:

* Awaiting any significant medical investigations relating to CPET absolute contraindications
* Hospitalisation within the last 4 weeks relating to CPET absolute contraindications
* Implantable cardiac devices e.g. pacemaker or implantable cardioverter defibrillator
* Unstable angina
* Unstable diabetes
* Left main coronary stenosis or its equivalent
* Known third degree heart block
* Unstable heart failure/New York Heart Association (NYHA) III or IV Heart Failure
* Acute aortic dissection, myocarditis, or pericarditis/endocarditis
* Suspected or known dissecting aneurysm
* Symptomatic severe aortic stenosis
* Acute deep vein thrombosis, pulmonary embolism or pulmonary infection
* Uncontrolled asthma
* Pulmonary oedema
* Respiratory failure
* Ambient O2 desaturation at rest <85%
* Resting tachycardia (>100bpm)
* Currently in atrial fibrillation
* Uncontrolled arrhythmia
* Resting systolic blood pressure >180 mmHg
* Resting diastolic blood pressure >100 mmHg
* Other conditions that prevent participants from completing study investigations (e.g. recent (last ~6 months) cardiac arrest)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with coronary heart disease currently enrolled in a Phase IV cardiac rehabilitation programme
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
V̇O2 peak agreement | Lab visit 30 minutes
  Agreement between V̇O2 peak recorded on a maximal CPET and V̇O2 peak estimated using VentriJect Seismofit

SECONDARY OUTCOMES:
V̇O2 peak repeatability | Lab visit 25 minutes
  Agreement between two V̇O2 peak estimations, recording using VentriJect Seismofit, taken 20 minutes apart

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Myers, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided